CLINICAL TRIAL: NCT02001610
Title: Clinical Trial of the Viability of LAB and Bifidobacteria From Acidophilus Pearls in Human Stool Samples
Brief Title: Acidophilus Pearls Fecal Recovery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Schwabe North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201300549; PS Project 00090915 (Other: University of Florida)
Record Dates: First submitted 2013-11-22; First posted 2013-12-05 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Survival of Probiotics During GI Transit; GI Symptoms
Keywords: microbiota; probiotics; fecal markers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hard shell gelatin capsules (Active Comparator): * Comparison delivery vehicle in the form of gelatin capsule
  * One capsule (containing at least 1 x 10^9 colony forming units) every morning for 12 days
  Interventions: Dietary Supplement: Hard shell gelatin capsules
- Acidophilus pearls (Experimental): * Encapsulated using patented process
  * One capsule (containing at least 1 x 10^9 colony forming units) every morning for 12 days
  Interventions: Dietary Supplement: Acidophilus pearls

INTERVENTIONS:
Dietary Supplement: Acidophilus pearls — * Acidophilus pearls are encapsulated using patented process
  * Subjects take one capsule (containing at least 1 x 10^9 colony forming units) every morning for 12 days
  Arms: Acidophilus pearls
Dietary Supplement: Hard shell gelatin capsules — * Hard-shelled gelatin capsule with same microbial formulation as pearl supplement
  * Subjects consume one capsule (containing at least 1 x 10^9 colony forming units) every morning for 12 days
  Arms: Hard shell gelatin capsules

SUMMARY:
Commercial probiotics can be delivered in numerous forms. The two most common delivery forms are similar to the two product formats to be tested. It has been demonstrated using in vitro testing that probiotic organisms that are unprotected from gastric exposure may not survive that exposure and therefore may not remain viable throughout the rest of the GIT. (Unpublished studies conducted at SNA research facility, February, 2010.) Similar in vitro testing of Acidophilus Pearls has demonstrated the probiotic organisms in an enteric capsule will survive gastric exposure. It is anticipated that this difference in in vitro gastric survivability will translate to improved digestive tract survivability that can be demonstrated using fecal recovery techniques.

The commercial product to be tested in this clinical trial has been in the market for over 17 years. However, it is not known what effect this commercial product has on the commensal probiotic population in the gut and particularly in the lower bowel where much of probiotic benefits are believed to be largely realized. Also, it is not known what effect the commercial product has on the total commensal microbiota or fecal pH. While commercial probiotic products have been largely aimed at benefits related to improved health, they also have the potential to change overall gut microbiota (probiotics as well as all others) composition and activities. Learning what happens to the overall gut microbiota can be a helpful step in establishing the potential health benefits of the probiotic class of organisms in the test products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Regular and predictable bowel movement pattern
* Willing to disclose OTC/prescription medications and dietary supplements taken during the study
* Willing to sign comprehensive informed consent form

Exclusion Criteria:

* Digestive disorders
* Use of prescribed medications that affect bowel function or microbiota (antibiotics, pain medications, laxatives)
* Use of dietary supplements/foods that can affect bowel function or microbiota
* Excessive alcohol use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in fecal survival of probiotics | Day 0 (before start of intervention), Day5-7 , Day 10-12 (end of intervention) and Day 17-19
  The investigators will measure survival of the probiotics in fecal samples.

SECONDARY OUTCOMES:
GI symptoms | Day 7-9 and day 10-12
  Change in GI symptoms using a weekly questionnaire.

OTHER OUTCOMES:
Fecal markers | Day 0 (before start of intervention), Day5-7 , Day 10-12 (end of intervention) and Day 17-19
  The investigators will measure fecal markers. This includes stool consistency on Bristol scale and pH.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Mai, PhD, Principal Investigator — University of Florida
Locations (1):
- Emerging Pathogens Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No